CLINICAL TRIAL: NCT01327521
Title: International Randomized Study of Transarterial Chemoembolization Versus CyberKnife for Recurrent Hepatocellular Carcinoma
Brief Title: Transarterial Chemoembolization vs CyberKnife for Recurrent Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Accrual below target levels
Sponsor: Albert Koong (Other)
Collaborators: Accuray Incorporated (Industry)
Responsible Party: Sponsor-Investigator, Albert Koong, Associate Professor of Radiation Oncology, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEP0030; ACCH001.0 (Other: Accuray Inc.); SU-05052010-5862 (Other: Stanford University)
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; Doxorubicin; Epirubicin; Fluorouracil; Mitomycin; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CyberKnife — Standard of Care
  Other Names: CK
Procedure: TACE — Standard of Care
  Other Names: Transcatheter arterial chemoembolization
Drug: CT Contrast — Standard of Care
  Other Names: contrast dye
Drug: doxorubicin — Standard of Care
  Other Names: Adriamycin; hydroxydaunorubicin
Drug: Epirubicin — Standard of Care
  Other Names: Ellence; Pharmorubicin; Epirubicin Ebewe
Drug: 5-fluorouracil — Standard of Care
  Other Names: 5-FU; f5U; Adrucil; Carac; Efudix; Efudex; Fluoroplex
Drug: Mitomycin C — Standard of Care
  Other Names: Mutamycin; MTC
Drug: Gemcitabine — Standard of Care
  Other Names: Gemzar
Drug: Cisplatin — Standard of Care
  Other Names: cisplatinum; cis-diamminedichloroplatinum(II); CDDP; Platinol; Platinol-AQ
Device: SMANCS — Standard of Care
  Other Names: styrene maleic acid neocarzinostatin; poppyseed oil

SUMMARY:
Primary Objective:

To compare the efficacy of TACE vs. CyberKnife SBRT in the treatment of locally recurrent HCC after initial TACE.

Secondary Objectives:

1. To determine the progression-free survival of TACE vs. CyberKnife SBRT
2. To determine the overall survival of TACE vs. CyberKnife SBRT for locally recurrent HCC
3. To determine the toxicities associated with TACE or CyberKnife SBRT for the treatment of recurrent HCC.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed hepatocellular carcinoma by one of the following:

  * Histopathology
  * One radiographic technique that confirms a lesion >=2 cm with arterial enhancement with washout on delayed phase
* Hepatic lesion in patients for whom surgical resection is not possible or would not result in an opportunity for cure
* Radiographic evidence of persistent, progressive or recurrent disease in an area previously treated with TACE. This evaluation should be determined after 6 weeks of initial TACE
* Multi-specialty evaluation whereby the recurrent liver lesion was deemed by both the attending radiation oncologist and interventional radiologist amenable to treatment by the respective modality

  * Eligible patients must undergo an IV contrast CT scan of the liver within 6 weeks of enrollment onto the study; a contrast enhanced liver MRI may be substituted for the IV contrast CT of the liver.
  * A recent serum AFP must also be obtained within 4 weeks of enrollment.
* Unifocal liver tumors not to exceed 7.5 cm in greatest axial dimension. Multifocal lesions will be restricted to lesions that can be treated within a single target volume within the same liver segment and to an aggregate of 7.5cm as long as the dose constraints to normal tissue can be met
* Eastern Clinical Oncology Group performance status 0, 1 or 2
* Patients with liver disease classified as Child Pugh class A/B; if Child's class B, score must be 8 or less
* Albumin >= 2.5 g/dL
* Total bilirubin <= 3 mg/dL
* INR <= 1.5
* Creatinine <= 2.0 mg/dL
* Age >= 18 years old
* Life expectancy>= 6 months
* Ability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior radiation for the recurrent liver tumors
* Prior radiotherapy to the upper abdomen
* Prior RFA to index lesion
* Liver transplant
* Tumors >= 7.5 cm in greatest axial dimension
* Portal vein thrombus
* Large varices within 2 cm of index lesion (seen on cross section imaging)
* Contraindication to receiving radiotherapy
* Active gastrointestinal bleed within 2 weeks of study enrollment
* Ascites refractory to medical therapy
* Women who are pregnant
* Administration of any systemic chemotherapy within the last 1 month
* Presence of multifocal lesions located in different lobes of the liver or extrahepatic metastases
* Participation in another concurrent SYSTEMIC treatment protocol
* Prior history of malignancy other than HCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Freedom from local progression at 6 months and 12 months | 6 months and 12 months

SECONDARY OUTCOMES:
Progression-free survival | at 6, 12 and 18 months
Overall survival | at 6, 12, 18 months and up to 3 years
Serum AFP levels | 1 month, 3 months, 6 months, 12 months and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert Koong, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States